CLINICAL TRIAL: NCT05959187
Title: A Single-center Randomized Controlled Study on the Effect of Pharmacogenomics Trial on Clinical Efficacy in Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-07-12
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Depressive Disorder; Pharmacogenomic Drug Interaction
Keywords: Depressive Disorder; Pharmacogenomic Drug Interaction
MeSH Terms: conditions — Depressive Disorder | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacogenomic testing group (Experimental): In the pharmacogenomic testing group, patients underwent collection of oral mucosal epithelial cells for common psychiatric drug gene testing, the clinical doctors were required to combine the patients' symptom characteristics with their own clinical experience and refer to the results of pharmacogenomic testing to guide drug treatment.
  Interventions: Diagnostic Test: pharmacogenomic testing
- Control (No Intervention): In the control group, patients did not undergo pharmacogenomic testing, and the clinical doctors were required to provide drug treatment based on their own diagnostic and therapeutic experience and the patients' symptom characteristics.

INTERVENTIONS:
Diagnostic Test: pharmacogenomic testing — Pharmacogenomic testing has emerged as a promising diagnostic tool, allowing clinicians to guide the selection and dosage of antidepressant medications. In theory, pharmacogenomic testing may provide improved drug selection and dosing strategies for patients with genetic alterations related to drug response
  Arms: Pharmacogenomic testing group

SUMMARY:
The purpose of this clinical trial is to explore the efficacy of drug therapy under the guidance of pharmacogenomics test in the treatment of patients with depression. The main questions to be answered in this study are:

1. Whether the drug treatment regimen under the guidance of pharmacogenomics test is beneficial to the rehabilitation of patients with depression.
2. Pharmacogenomics tests whether it can reduce adverse drug reactions during treatment, and be evaluated by the scale before and after treatment.

The researchers will compare the pharmacogenomics test group with the healthy control group to see the effect of drug therapy under the guidance of pharmacogenomics test on the efficacy of patients with depression.

DETAILED DESCRIPTION:
Drug treatment of mental disorders is often seriously hindered by huge differences in individual drug responses or drug side effects, which are closely related to genetic factors. Pharmacogenomics testing can help clinicians to provide better drug choices for patients. In this study, a single center randomized controlled design was used, including 300 cases in the drug gene detection group and 300 cases in the healthy control group. Hamilton Depression scale (HAMD) and side effects scale (TESS) were used to evaluate the efficacy of pharmacogenomics test in the treatment of depression before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosis of depressive disorder based on DSM-V criteria by two or more senior psychiatrists; 2) Hamilton Depression Scale (HAMD) score more than 14; 3) Age between 14 and 75 years; 4) Completed at least middle school education or higher and capable of completing the assessment scales; 5) Good compliance with medication treatment.

Exclusion Criteria:

1) Presence of mental retardation or significant medical history of other major physical illnesses (including a history of cranial trauma or infection, intracranial tumors, cerebrovascular diseases, epilepsy, etc.); 2) History of benzodiazepine sedative-hypnotic drug, alcohol, or other substance abuse; 3) History of electroconvulsive therapy; 4) Pregnancy or lactation.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
remission | Change the percentage of remission from baseline in the fourth week of intervention
  remission, defined as a HAMD-24 score of 7 or less after treatment.
response | Change the percentage of response from baseline in the fourth week of intervention
  response, defined as a HAMD-24 score at least 50% decrease from the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Lin, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China